CLINICAL TRIAL: NCT02809677
Title: Treating Caregiver Depression to Improve Childhood Asthma: Impact and Mediators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University at Buffalo (Other)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 022014-069; 1R01HL123609-01A1 (NIH)
Record Dates: First submitted 2016-04-11; First posted 2016-06-22 (Estimated); Results first posted 2022-02-15 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Asthma; Major Depressive Disorder
MeSH Terms: conditions — Asthma; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Study followed caregivers and children for up to 12 months. They were given the option of algorithm-based antidepressant therapy using a variety of standard treatments. However, they could also receive medication or psychotherapy outside of the study, or decline all treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Non-Interventional Longitudinal Study (Other): This is a 52 week non-placebo controlled and non-randomized clinical research study to see whether treating Major Depressive Disorder (MDD) in caregivers of children with asthma will improve asthma outcomes in children. Caregivers may choose to receive an antidepressant medication that is considered standard medical care for MDD, or may opt out of antidepressant treatment. No treatment is withheld from participants and no placebos are used, thus there is no active intervention in this study.
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — This is a 52 week non-placebo controlled and non-randomized clinical research study to see whether treating Major Depressive Disorder (MDD) in caregivers of children with asthma will improve asthma outcomes in children. Caregivers may choose to receive an antidepressant medication that is considered standard medical care for MDD, or may opt out of antidepressant treatment. No treatment is withheld from participants and no placebos are used, thus there is no active intervention in this study.

SUMMARY:
The investigators propose a one-year, repeated measures, within-subject design to examine the impact of improved caregiver depression on child asthma outcomes. A cross-lagged panel modeling (CLPM) for longitudinal data will be fit using a maximum likelihood structural equation model (SEM) in order to explore longitudinal mediation between asthma outcomes (asthma control, spirometry, quality of life (QOL)) and depressive symptoms. CLPM will test whether caregiver improvement preceded child asthma improvement, and SEM will test whether improved adherence and/or decreased child anxiety/depression mediated the effect. The investigators considered a randomized control trial, but it would not be ethically acceptable to withhold medication from caregivers diagnosed with Major Depressive Disorder (MDD) for the proposed one-year duration of the study. It is unlikely that potential participants in the study would find this acceptable. Furthermore a controlled design is not necessary since the investigators are not testing the efficacy of antidepressants for depression, but rather the impact of improvement on caregiver depression on the child.

DETAILED DESCRIPTION:
Caregiver will be consented for his/her and the child's participation. The child will assent to participate before study procedures begin. The proposed study will last 52 weeks and consist of study visits every 4 weeks (14 visits total).

Screening (roughly 5 mins):

2 item Self-Report Screening Tool for Depression (2-SRSD) This tool will be used to help screen caregivers for the study.

This screening will only be performed in the clinic. Additional screening will be performed at the Baseline visit including:

* Obtaining demographic information
* Physical exam,
* Medical and psychiatric history
* Physical health assessments
* Urine Pregnancy Test for women of childbearing potential
* Mood assessments

The baseline visit is described below:

Baseline (approx 3 hrs):

The following assessments will be given to the Caregiver only:

1. Structured Clinical Interview for DSM V (SCID)
2. Urine Pregnancy Test (UPT) for women of child bearing potential
3. Hamilton Rating Scale for Depression (HRSD)
4. Quick Inventory of Depressive Symptomatology Self Report (QIDS-SR)
5. State Trait Anxiety Inventory (STAI)
6. Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQOL)
7. Psychobiology of Recovery in Depression III Somatic Symptom Scale (PRD-III)

The following assessments will be given to the child:

1. Composite Asthma Severity Index (CASI)
2. Children's Depression Inventory (CDI)
3. Screen for Child Anxiety Related Disorders (SCARED)
4. Pediatric Asthma Quality of life Questionnaire (PAQOL)
5. Asthma Control Test/Childhood Asthma Control Test (ACT/cACT) (which version is given will be determined by the child's age)
6. Spirometry measurement
7. Perceived Stress Scale (PSS)
8. Relatedness Scale

The following assessments will be given to both the caregiver AND the child:

1. Childhood Asthma Management Program Continuation Study Medication Adherence Interview (CAMPCS)

Weeks 4-48 (visits every 4 weeks, each approx 2 hours):

Caregiver only:

HRSD, QIDS-SR, STAI, PACQOL, PRD-III, UPT

Child only:

CASI, CDI, SCARED, PAQOL, ACT/cACT, Spirometry, PSS, Relatedness Scale

Both caregiver AND child:

CAMPCS

Week 52 (approx 2.5 hrs):

Caregiver only:

HRSD, QIDS-SR, STAI, PACQOL, PRD-III, UPT

Child only:

CASI, CDI, SCARED, PAQOL, ACT/cACT, Spirometry, PSS, Relatedness Scale

Both caregiver AND child:

CAMPCS, Debriefing interview

Electrocardiograms (ECG) and blood tests may be collected during this study as is clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver: Male or female, ages 18 to 70, primary asthma caregiver of the child, currently meeting criteria for Major Depressive Disorder (MDD) (based on depression symptoms for at least 2 weeks and causing clinically significant distress or impairment in social, occupational, or other important areas of functioning) based on a Structured Clinical Interview for DSM-4 (SCID) interview.
* Child: Male or female, ages 7-17 years who have a diagnosis of persistent asthma as classified by either of the following criteria:
* A. requirement for treatment with daily controller medication; or
* B. symptoms of persistent asthma in children not on a daily controller medication:
* 1. Daytime symptoms two or more days per week; or
* 2. Rescue bronchodilator use two or more times per week; or
* 3. Nocturnal symptoms two or more nights per month; or
* 4. Two or more oral steroid bursts in the last year.

Exclusion Criteria:

* Caregiver: Severe cognitive impairment that could impair their ability to provide informed consent; member of a vulnerable population (incarcerated, pregnant or breastfeeding women); women of childbearing age who will not use acceptable methods of birth control or abstinence during the study; severe psychiatric disorder in addition to MDD that should be a primary focus of treatment (e.g. severe and disabling eating or anxiety disorders); treatment refractory depression defined as failing ≥ 3 adequate trials of antidepressants (≥ 4 weeks at a therapeutic dose); electroconvulsive therapy or repeated transcranial magnetic stimulation during the current episode; depression as part of bipolar disorder or schizophrenia or schizoaffective disorder, or current depression secondary to substances or general medical condition, or with psychotic features or accompanied by severe obsessive compulsive disorder (OCD), or high risk for suicide defined by multiple recent suicide attempts (> 2 in the past year) or any attempt in the past month, or current suicidal ideation with a well-formed plan or intent.
* Child: Severe cognitive impairment that could impair their ability to provide informed consent; high risk for suicide defined by multiple recent suicide attempts (> 2 in the past year) or any attempt in the past month, or current suicidal ideation with a well-formed plan or intent; severe or life-threatening medical illness, such as other serious cardiopulmonary conditions (e.g. congenital heart disease, cystic fibrosis, alpha-1-antitrypsin disease) or cancer, which would confound the assessment of asthma, anxiety, depression or quality of life; severe psychiatric illness, such as autism, bipolar disorder, schizophrenia or current drug/alcohol abuse/dependence. If an eligible caregiver presents with more than one child meeting inclusion criteria for the study, only one child, randomly selected, will be enrolled.

Ages: 7 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edson S Brown, M.D., PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center Psychoneuroendocrine Research Program, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gwak DY, Tea JC, Fatima FN, Palka JM, Lehman H, Khan DA, Zhou H, Wood BL, Miller BD, Brown ES. Contribution of caregiver and child anxiety and depressive symptoms to child asthma-related quality of life. Ann Allergy Asthma Immunol. 2024 Sep;133(3):295-301. doi: 10.1016/j.anai.2024.02.026. Epub 2024 Mar 6. PMID 38458318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants included depressed caregivers and children with asthma, being treated at UT Southwestern (Dallas) and SUNY-Buffalo medical centers.
Groups:
- Caregiver Child Dyad: Caregivers may choose to receive an antidepressant medication that is considered standard medical care for MDD, or may opt out of antidepressant treatment. No treatment is withheld from participants and no placebos are used, thus there is no active intervention in this study.
Period: Overall Study
Arm/Group | Caregiver Child Dyad
Started | 205
Completed | 197
Not Completed | 8
Not completed — Withdrawal by Subject | 8

BASELINE CHARACTERISTICS:
Groups:
- Caregiver Child Dyad: This is a 52 week non-placebo controlled and non-randomized clinical research study to see whether treating Major Depressive Disorder (MDD) in caregivers of children with asthma will improve asthma outcomes in children. Caregivers may choose to receive an antidepressant medication that is considered standard medical care for MDD, or may opt out of antidepressant treatment. No treatment is withheld from participants and no placebos are used, thus there is no active intervention in this study.
Arm/Group | Caregiver Child Dyad
Number analyzed (Participants) | 205
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Caregiver | 38.62 (7.95)
  Child | 11.31 (2.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Caregiver: Female | 201
  Caregiver: Male | 4
  Child: Female | 111
  Child: Male | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Caregiver: Hispanic or Latino | 65
  Caregiver: Not Hispanic or Latino | 134
  Caregiver: Unknown or Not Reported | 6
  Child: Hispanic or Latino | 65
  Child: Not Hispanic or Latino | 132
  Child: Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Caregiver: American Indian or Alaska Native | 4
  Caregiver: Asian | 1
  Caregiver: Native Hawaiian or Other Pacific Islander | 0
  Caregiver: Black or African American | 107
  Caregiver: White | 81
  Caregiver: More than one race | 12
  Caregiver: Unknown or Not Reported | 0
  Child: American Indian or Alaska Native | 2
  Child: Asian | 1
  Child: Native Hawaiian or Other Pacific Islander | 0
  Child: Black or African American | 116
  Child: White | 71
  Child: More than one race | 12
  Child: Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 205
Asthma Control Test (ACT) [Mean (Standard Deviation); unit: units on a scale] — ACT is a patient self-administered tool for identifying those with poorly controlled asthma. It is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled). The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
  units on a scale | 17.78 (4.89)
Childhood Asthma Control Test (cACT) [Mean (Standard Deviation); unit: units on a scale] — Childhood Asthma Control Test (C-ACT) is well validated for use among children aged 4-11 years comprised of 3 parent-reported and 4 child-reported items. Possible scores range from 0 to 12, with higher scores indicating better asthma control.
  units on a scale | 17.47 (4.64)
Hamilton Rating Scale for Depression (HRSD) [Mean (Standard Deviation); unit: units on a scale] — Caregiver depressive symptoms were assessed with the Hamilton Rating Scale for Depression (HRSD) which is a 17 item scale. Range: 0-53 Normal: 0-7 Mild: 8 - 13 Moderate 14 - 18 Severe: 19-22 Very severe > 22
  units on a scale | 17.95 (4.79)
Children's Depression Inventory-Short Form (CDI-SF) [Mean (Standard Deviation); unit: units on a scale] — 10-item CDI-S asks respondents to rate the severity of different symptoms of depression. Each item consists of three statements graded in order of increasing severity from 0 to 2. The item scores are combined into a total depression score, which ranges from 0 to 54, where higher scores indicate more depressive symptomatology (worse outcome).
  units on a scale | 9.50 (6.36)
Spirometry (FEV1%) [Mean (Standard Deviation); unit: Percentage of FEV1 % predicted] | 73.79 (38.11)
Medication Adherence (prescribed inhalers) [Mean (Standard Deviation); unit: Percentage of prescribed puffs] — Medication adherence was assessed as a percent of prescribed puffs children were adherent to at the Baseline assessment
  Percentage of prescribed puffs | 72.17 (31.45)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression (HRS-D) Change Scores
Description: Change from Baseline in the caregiver's depression scores, as assessed by Hamilton Rating Scale for Depression (HRS-D). HRSD is a 17 item scale. Range: 0-53 Normal: 0-7 Mild: 8 - 13 Moderate 14 - 18 Severe: 19-22 Very severe > 22
Time Frame: From date of Baseline until the date of first documented progression, assessed up to 52 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Child Dyad
Number analyzed (Participants) | 197
units on a scale | -8.39 (7.37)

2. Primary Outcome: Asthma Control Test (ACT) Change Scores
Description: Change from Baseline in the child's asthma control scores, as indicated by increased Asthma Control Test (ACT) scores. ACT is a patient self-administered tool for identifying those with poorly controlled asthma. It is a 5-point scale (for symptoms and activities: 1=all the time to 5= not at all; for asthma control rating: 1=not controlled at all to 5=completely controlled). The scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Time Frame: From date of Baseline until the date of first documented progression, assessed up to 52 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Child Dyad
Number analyzed (Participants) | 197
units on a scale | 2.71 (4.80)

3. Primary Outcome: Composite Asthma Severity Index (CASI) Change Scores
Description: Change from Baseline in the child's asthma control scores, as indicated by decreased Composite Asthma Severity Index (CASI) scores. The Composite Asthma Severity Index (CASI) is a comprehensive severity scale combining multiple facets of asthma severity: impairment, risk, and treatment and ranges from 0 to 20 points, with higher scores indicating higher levels of severity.
Time Frame: From date of Baseline until the date of first documented progression, assessed up to 52 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Child Dyad
Number analyzed (Participants) | 197
units on a scale | -1.43 (2.74)

4. Primary Outcome: Quick Inventory of Depressive Symptomology - Self Report (QIDS-SR) Change Scores
Description: Change from Baseline in the caregiver's depression scores, as assessed by Quick Inventory of Depressive Symptomology - Self Report (QIDS-SR). The QIDS-SR is a validated 16-item self-report scale that assesses depressive symptom severity. Total QIDS-SR scores range from 0 to 27. Scores of ≤ 7 are considered normal, 8-12 suggest mild depressive symptoms, 13-16 moderate depressive symptoms, 17-20 moderate to severe depressive symptoms, and ≥ 21 severe depression.
Time Frame: From date of Baseline until the date of first documented progression, assessed up to 52 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Child Dyad
Number analyzed (Participants) | 197
units on a scale | -7.12 (5.55)

5. Primary Outcome: Childhood Asthma Control Test (cACT) Change Scores
Description: Change from Baseline in the child's asthma control scores, as indicated by increased Childhood Asthma Control Test (cACT) scores. Childhood Asthma Control Test (C-ACT) is well validated for use among children aged 4-11 years comprised of 3 parent-reported and 4 child-reported items. Possible scores range from 0 to 12, with higher scores indicating better asthma control.
Time Frame: From date of Baseline until the date of first documented progression, assessed up to 52 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Child Dyad
Number analyzed (Participants) | 197
units on a scale | 0.93 (2.63)

6. Secondary Outcome: Number of Unscheduled Asthma-related Service Utilization Visits (Child)
Description: Number of unscheduled asthma-related service utilization visits (i.e., clinic visits, ER visits, and hospitalizations) for the child participant at 52 weeks.
Time Frame: 52 weeks.
Measure: Number; unit: Visitis
Arm/Group | Caregiver Child Dyad
Number analyzed (Participants) | 197
Visitis
  Unscheduled Clinic Visits | 70
  ER Visits | 48
  Hospitalizations | 17

7. Secondary Outcome: Pediatric Asthma Quality of Life Questionnaire (PAQOL) Change Scores
Description: Change from Baseline in child's quality of life scores on the Pediatric Asthma Quality of Life Questionnaire. Pediatric Asthma Quality of Life Questionnaire (PAQOL) measures problems that children experience as a result of their asthma. It has 23 questions in 3 domains (symptoms, activity limitation and emotional function). The activity domain contains 3 'patient-specific' questions. Children are asked to think about how they have been during the previous week and to respond to each of the 23 questions on a 7-point scale (7 = not bothered at all - 1 = extremely bothered). Higher scores indicate better levels of functioning. This scale has proved a valid and reliable measure of asthma-specific quality of life in adolescents. Mean scores are reported, and range from 1 to 7. Higher score indicating higher quality of life.
Time Frame: From date of Baseline until the date of first documented progression, assessed up to 52 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregiver Child Dyad
Number analyzed (Participants) | 197
units on a scale | 0.85 (1.92)

8. Secondary Outcome: Percent Change in Medication Adherence (Prescribed Inhalers)
Description: Percent change in Medication Adherence (prescribed inhalers) was assessed by responses to items 4 (i.e., "The days that you took your controller medication in the last 7 days, about how much did you usually take each day?") and 5 (i.e., "How many days in the past 7 days did you take this controller medication?") from Childhood Asthma Management Program Continuation Study (CAMPCS) multiplied to determine how many puffs of the inhaled controller therapy were taken in the prior seven days. Following this, the product of items 4 and 5 was divided by the prescribed number of puffs per week (taken from RedCap).
Time Frame: Baseline, 52 weeks (1 year).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Caregiver Child Dyad
Number analyzed (Participants) | 197
percent change | 13 (41)

ADVERSE EVENTS:
Time Frame: 4 years, 4 months
Description: Definitions do not differ from clinicaltrials.gov definitions.
Arm/Group | Caregiver Child Dyad
All-Cause Mortality (participants affected / at risk) | 0/205
Serious Adverse Events (participants affected / at risk) | 0/205
Other Adverse Events (participants affected / at risk) | 46/205
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caregiver Child Dyad (N=205)
Headache (General disorders) | 11 (11)
Infections (General disorders) | 21 (21)
Nausea and/or vomiting (Gastrointestinal disorders) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT02809677/Prot_SAP_000.pdf